CLINICAL TRIAL: NCT04361981
Title: National Cohort Study to Assess the Influence of COVID-19 Infection in Thromboembolic Venous Disease:
Brief Title: Influence of COVID-19 Infection in Thromboembolic Venous Disease: National Cohort Study
Acronym: TVP-COVID-RIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sociedad Espanola de Angiologia y Cirugia Vascular (Network)
Responsible Party: Sponsor
Other Study IDs: RIV-R3
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: COVID-19 infection patients with a Deep Venous Disease event
  Interventions: Other: Deep Venous Disease Diagnostic

INTERVENTIONS:
Other: Deep Venous Disease Diagnostic — Clinical and/or echographic diagnosis of Deep Venous Disease in a patient with COVID-19 infection

SUMMARY:
There is an urgent need to understand the outcomes of COVID-19 infected patients regarding the thromboembolic venous disease. Capturing real-world data and sharing Spanish national experience will inform the management of this complex group of patients, improving their clinical care.

Interventions are needed to reduce both the incidence and severity of COVID-19. Although it shares characteristics with other similar viruses that also arose in outbreaks, the physiological mechanisms of the virus and its responses on the host are not yet fully known. There are indications that the clinical picture of this disease is in a procoagulant state, with possible increase in episodes of thromboembolic disease. This study aims to analyze the influence of COVID-19 on the incidence of deep vein thrombosis (DVT) in lower and upper limbs, and the variation in the clinical presentation of COVID-19, as well as to provide new evidence applicable to the clinical management of these patients and the establishment of prognostic factors that help early take therapeutic decisions.

To this end, an observational, multicenter, national cohorts study will be carried out, sponsored by the Spanish Society of Angiology and Vascular Surgery (SEACV) and the Spanish Chapter of Phlebology and Linfology through its Vascular Research Network (RIV), which will collect demographic variables, comorability, concomitant treatment, analytical status and complementary and ultrasound diagnostic tests, parameters of clinical evolution, therapeutic and complications and mortality to 30 days. All national centers you wish to participate through a secure server that will be accessed through the SEACV and CEFyL website.

The global community has recognised that rapid dissemination and completion of studies in COVID-19 infected patients is a high priority, so we encourage all stakeholders (local investigators, ethics committees, IRBs) to work as quickly as possible to approve this project.

This investigator-led, non-commercial, non-interventional study is extremely low risk, or even zero risk. This study does not collect any patient identifiable information (including no dates) and data will not be analysed at hospital-level.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years) considered as a case of COVID-19 disease with suspected DVT in lower and/or upper limbs: (i) A laboratory test confirming COVID-19 infection or (ii) a clinical diagnosis of COVID-19 infection (without any testing) is considered.

  - Suspected DVT:
* Patients with clinical data of suspected DVT
* and/or patients with analytical data on suspected DVT
* and/or patients with ultrasound data of suspected DVT

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COVID-19 infection who suffer from deep venous disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Deep Venous Disease Incidence | 30 days
  Incidence of Deep Venous Disease events in patients with COVID-19 infection

SECONDARY OUTCOMES:
30-days mortality | 30 days
  30-days mortality in COVID-19 infection patients with a Deep Venous Disease event
ICU admission | 30 days
  Rate of ICU admission in COVID-19 infection patients with a Deep Venous Disease event
Anticoagulant treatment | 30days
  Type of anticoagulant treatment in COVID-19 infection patients with a Deep Venous Disease event

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin De Haro, MD, Study Chair — Hospital Universitario Getafe. Red de Investigacion Vascular
Locations (1):
- Red de Investigacion Vascular (SEACV), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided